CLINICAL TRIAL: NCT00954902
Title: Development of a Dynamic Model of Inflammation for Studying the Anti-inflammatory Effects of Culinary Spices in Human Participants
Brief Title: Effects of Antioxidants on Cardiovascular Risk Measures (Spice Study)
Acronym: Spice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Principal Investigator, Sheila G West, Professor of Biobehavioral Health, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: G264
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Cardiovascular; Psychological Stress
Keywords: Spice; responses to stress; Inflammatory
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- No spice, no stress (Sham Comparator): Subject are given placebo capsules and told they contain an antioxidant concentrate
  Interventions: Other: Placebo antioxidant concentrate
- No Spice, Stress (Sham Comparator): Subjects are given placebo capsules and told they are receiving an equivalent amount of an antioxidant concentrate.
  Interventions: Behavioral: Trier Psychological Stressor; Other: Placebo antioxidant concentrate
- Spice, no stress (Experimental)
  Interventions: Dietary Supplement: High Antioxidant Spice Blend
- Spice and Stress (Experimental)
  Interventions: Dietary Supplement: High Antioxidant Spice Blend; Behavioral: Trier Psychological Stressor

INTERVENTIONS:
Dietary Supplement: High Antioxidant Spice Blend — 14.5 g spice blend incorporated into a delivery meal including: cloves, cinnamon, oregano, rosemary, ginger, black pepper, paprika, garlic powder, and turmeric.
  Arms: Spice and Stress; Spice, no stress
Behavioral: Trier Psychological Stressor — This is a psychological stressor that is used to invoked stress responses in human subjects. Subjects are told they are taped and evaluated and deliver the speech in front of a trained panel of judges.
  Arms: No Spice, Stress; Spice and Stress
Other: Placebo antioxidant concentrate — Placebo capsules
  Arms: No Spice, Stress; No spice, no stress

SUMMARY:
The purpose of this study is to assess whether feeding highly antioxidant spices of providing these same antioxidants as capsules is able to affect cardiovascular risk measures. Because this is a new area of research, the investigators will use many measures to assess this question including blood markers, tests of blood vessel health, measures of blood pressure responses, measures of clotting activity, and other inflammation measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65
* BMI 25-40
* Non tobacco user
* Resting BP < 160/100
* Fasting Glucose < 126 mg/dL

Exclusion Criteria:

* Tobacco use
* Use of female hormones
* Breastfeeding or planning to become pregnant during the study
* Use of lipid-lowering or blood pressure medications
* Chronic Inflammatory Disease or osteoarthritis requiring regular use of medication
* Chronic use of any form of anti-inflammatory or anti-psychotic drugs
* Use of daily aspirin or supplements (except stable dose of calcium)
* History of heart attack or stroke, renal or hepatic disease, implanted medical devices, gastrointestinal disease
* Allergy or intolerance to any study foods
* Injury to fingers or arms that would interfere with vascular and blood pressure measurements
* Inability to comply with study protocol
* Allergy to adhesives or latex
* Aerobic exercise exceeding 2 hours per week

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
IL-6 response to psychological stress at time points equal to and greater than 90 minutes post task | At baseline and intervals up to 2 hours following the stressor and 3.5 hours following the meal

SECONDARY OUTCOMES:
Serum/plasma changes in antioxidant activity and their relationship to inflammation outcomes | At baseline and intervals up to 2 hours following the stressor and 3.5 hours following the meal
Endothelial function measured by endopat | At baseline and 3.5 hours following the meal
Platelet function measured by PFA-100 | At baseline and specified intervals up to 2 hours following the stressor and 3.5 hours following the meal

CONTACTS AND LOCATIONS:
Overall Officials: Sheila G. West, PhD, Principal Investigator — Penn State; Ann C. Skulas-Ray, B.S., Principal Investigator — Penn State; Penny M. Kris-Etherton, PhD, RD, Principal Investigator — Penn State
Locations (1):
- Penn State GCRC, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] McCrea CE, West SG, Kris-Etherton PM, Lambert JD, Gaugler TL, Teeter DL, Sauder KA, Gu Y, Glisan SL, Skulas-Ray AC. Effects of culinary spices and psychological stress on postprandial lipemia and lipase activity: results of a randomized crossover study and in vitro experiments. J Transl Med. 2015 Jan 16;13:7. doi: 10.1186/s12967-014-0360-5. PMID 25592751